CLINICAL TRIAL: NCT07089706
Title: A Phase 3b/4, Open-label Study to Evaluate the Immunogenicity and Safety of mRNA-1283 COVID-19 Variant-containing Vaccine Formulations
Brief Title: A Study to Evaluate the Immunogenicity and Safety of mRNA-1283 COVID-19 Variant-containing Formulations
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: mRNA-1283-P401
Record Dates: First submitted 2025-07-21; First posted 2025-07-28 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: COVID-19
Keywords: mRNA-1283; mRNA-1283 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Coronavirus Infections; Virus Diseases; mNEXSPIKE®; COVID-19; COVID-19 vaccine; Moderna
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Virus Diseases

STUDY DESIGN:
Intervention Model Description: This is a Phase 3b/4 open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mRNA-1283.251 Variant-containing Formulation (Experimental): Participants will receive an intramuscular (IM) injection of a mRNA-1283.251 variant-containing formulation.
  Interventions: Biological: mRNA-1283.251 Variant-containing Formulation

INTERVENTIONS:
Biological: mRNA-1283.251 Variant-containing Formulation — Sterile liquid for injection
  Other Names: mNEXSPIKE®

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of the recommended variant-containing formulations of mRNA-1283 COVID-19 vaccine (mNEXSPIKE®) within the current epidemiological environment.

DETAILED DESCRIPTION:
This study uses a master protocol with a generic study design to allow flexibility in evaluating immunogenicity of variant-containing formulations of the mRNA-1283 COVID-19 vaccine. As different variant-containing vaccine formulations will be evaluated, each study intervention (for example, updated mRNA-1283 COVID-19 vaccine) will be described in the subprotocol. For each evaluation of an updated variant vaccine, a new subprotocol will be generated.

Subprotocol 01 is a single arm study to evaluate immunogenicity and safety of mRNA-1283 (COVID-19 vaccine) 2025-2026 formula in individuals aged ≥65 years and ≥12 to <65 years with at least 1 underlying condition that puts them at high risk for severe outcomes from COVID-19.

The study included Parts A and B. Part A enrollment was discontinued due to addition of Part B to evaluate the safety and immunogenicity of variant-containing mRNA-1283 using a hypothesis driven study endpoint with reactogenicity data collection and longer safety follow up in Part B.

ELIGIBILITY:
Inclusion Criteria:

Subprotocol 1:

* ≥65 years of age at the time of signing the informed consent or ≥12 to <65 years of age at the time of signing the informed consent with at least 1 risk factor for severe outcomes from COVID-19.
* Investigator's assessment that the participant understands and is willing and physically able to comply with protocol-mandated follow-up, including all procedures.
* Participants who are assigned female at birth or could become pregnant:

  i) Has a negative pregnancy test at the Screening Visit and on the day of vaccination prior to vaccine dose being administered on Day 1.

ii) Has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first dose (Day 1).

iii) Has agreed to continue adequate contraception through 28 days following vaccine administration.

Exclusion Criteria:

Subprotocol 1:

* History of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 6 months prior to enrollment.
* Acutely ill or febrile (temperature ≥38.0°Celsius/≥100.4°Fahrenheit) within 72 hours prior to or at the Screening Visit or Day 1. Participants meeting this criterion may be rescheduled within the Screening window and will retain their initially assigned participant number.
* History of a diagnosis or condition that, in the judgment of the Investigator, is clinically unstable or may affect participant safety, assessment of study endpoints, assessment of immune response, or adherence to study procedures.
* Receipt of the COVID-19 vaccine within 6 months prior to enrollment.
* Receipt of any licensed non-COVID-19 vaccine within 28 days before or planned receipt within 28 days after the study intervention, except an influenza vaccine, which may be given 14 days before or after receipt of the study intervention.
* Receipt of systemic immunosuppressants for >14 days in total, within 180 days prior to Screening Visit (for corticosteroids ≥10 milligrams [mg]/day of prednisone equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study.
* Receipt of systemic immunoglobulins, long-acting biological therapies that affect immune responses (for example, infliximab) or blood products within 90 days prior to the Screening Visit or plans to receive them during the study.
* History of anaphylaxis or severe hypersensitivity reaction requiring medical intervention after receipt of any mRNA vaccine or therapeutic or any components of an mRNA vaccine or therapeutic.
* Has donated ≥450 milliliters (mL) of blood products within 28 days prior to the Screening Visit or plans to donate blood products within 28 days after the study injection.

Note: Other protocol-specified inclusion and exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 832 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-05-11 (Estimated); Study Completion 2026-05-11 (Estimated)

PRIMARY OUTCOMES:
Subprotocol 1: Part A - Geometric Mean (GM) Value of Neutralizing Antibody (nAb) Against Vaccine-matched COVID-19 Variants | Day 29
Subprotocol 1: Part A - Geometric Mean Fold Rise (GMFR) of nAb Against Vaccine-matched COVID-19 Variants | Baseline to Day 29
Subprotocol 1: Part B - GMFR of nAb Against Vaccine-matched COVID-19 Variants | Baseline to Day 29
Subprotocol 1: Part A - Seroresponse Rate (SRR) of nAb Against Vaccine-matched COVID-19 Variants | Baseline to Day 29

SECONDARY OUTCOMES:
Subprotocol 1: Part A - Number of Participants with Unsolicited Adverse Events (AEs), Serious Adverse Events (SAEs), AEs of Special Interests (AESIs), and AEs Leading to Study Withdrawal | Day 1 through Day 29
Subprotocol 1: Part B - Number of Participants with Unsolicited AEs | Day 1 through Day 29
Subprotocol 1: Part B - Number of Participants with SAEs, AESIs, and AEs Leading to Study Withdrawal | Day 1 through Day 181
Subprotocol 1: Part B - Geometric Mean Ratio (GMR) of nAb Against Vaccine-matched COVID-19 Variants Between Participants Aged ≥12 to <65 Years and Those Aged ≥65 Years | Day 29
Subprotocol 1: Part B - Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs) | 7 days post vaccination

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - DelRicht Research-Atlanta, Atlanta, Georgia
  - DelRicht Research-Baton Rouge, Baton Rouge, Louisiana
  - DelRicht Research-New Orleans, New Orleans, Louisiana
  - DelRicht Research-Gulfport, Gulfport, Mississippi
  - DelRicht Research-Tulsa, Tulsa, Oklahoma